CLINICAL TRIAL: NCT06833086
Title: Evaluation of Influence of Thoracic Paravertebral Block on Atrioventricular Conduction
Brief Title: Influence of Thoracic Paravertebral Block on Atrioventricular Conduction
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Prof., Medical University of Gdansk
Other Study IDs: KB/35/2025
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Conduction Abnormalities; Paravertebral Anesthesia
Keywords: P wave; PR interval; PQ interval; P wave dispersion; Paravertebral block; Atrioventricular conduction; Ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- L - paravertebral block left: 30 woman above 18 years of age qualified for elective breast surgery on the left side of the body
  Interventions: Procedure: Paravertebral block (ropivacaine) left
- P - paravertebral block right: 30 woman above 18 years of age qualified for elective breast surgery on the right side of the body
  Interventions: Procedure: Paravertebral block (ropivacaine) right

INTERVENTIONS:
Procedure: Paravertebral block (ropivacaine) left — Paravertebral block at the level of 3rd thoracic intervertebral space on the left side. 0.5% Ropivacaine 0.3 ml·kg-1, not exceeding 30 ml, based on ideal body weight in obese patients
  Groups: L - paravertebral block left
Procedure: Paravertebral block (ropivacaine) right — Paravertebral block at the level of 3rd thoracic intervertebral space on the right side. 0.5% Ropivacaine 0.3 ml·kg-1, not exceeding 30 ml, based on ideal body weight in obese patients
  Groups: P - paravertebral block right

SUMMARY:
The aim of the study is to assess the changes in electrical activity of heart atria and in atrioventricular conduction induced by anaesthetic thoracic paravertebral blockade, depending on site on which blockade was performed.

Researchers will retrospectively compare ECG recordings of patients that undergone unilateral paravertebral blockade at T3 level with 0.5% ropivacaine. The investigation will include measurement of P wave and PR interval, and subsequent statystical analysis.

DETAILED DESCRIPTION:
Paravertebral blockade (PVB), the injection of local anaesthetic into the paravertebral space located along the vertebral column, temporarily impair the transmission in nerve fibers located in this space. Although PVB is usually used primarily with the intention of achieving block of the thoracic wall pain sensation, the paravertebral space contains not only motoric and sensory nerves, but also autonomic nerve fibers. Achieving the blockade at top four thoracic levels of paravertebral space may affect, among the others, the function of preganglionic sympathetic fibers, forming cardiac nerves, and affecting the heart function in various ways.

The assessment of electrocardiographical phenomena representing the depolarisation of the atria (P wave) and the propagation of the depolarisation by the atrioventricular node and bundle (PQ/PR interval) allows to detect the abnormalities related to proability of occurrence of supraventricular arrythmias and conduction blocks, including the life-threatening arrythmias.

The design of the study assume to retrospective re-analyse the electrocardiographical data achieved in the "Influence of Thoracic Paravertebral Block on Cardiac Repolarization" study (registred in Clinicaltrials.gov under ID NCT05822076), focused changes in heart repolarisation represented mainly by electrocardiographical QT interval and T wave dispersion.

The population of primary investigation was 60 women above 18 years of age scheduled to elective breast surgery in combined regional and general anaesthesia will be enrolled to study, divided in two groups depending of the side of operation. Participants underwent the ultrasound-guided paravertebral block with single injection of 0.5% ropivacaine (0.3 ml·kg-1, not exceeding 30 ml, based on ideal body weight in obese patients) without adjuvants. Before injection (T0) and after confirmation of sufficient sensory block area covering 1st to 4th thoracic dermatomes (T1), 12-lead electrocardiogram (ECG) will be recorded using a Holter device. First examination of sensory block distribution was performed 6 minutes after injection, with subsequent examinations if needed - every minute up to 15 minutes. No sedative premedication, general anaesthesia induction or additional medications (except of neutral saline maintaining intravenous access) were administered until completions of ECG recording. Both T0 and T1 electrocardiogram will be preceded by rest in supine position for at least 5 minutes, without any medical procedures other than monitoring.

As part of the retrospective analysis of ECG recordings obtained from the primary study, repeated measurements will be performed to assess the length of the P wave and the PQ interval at time points T0 and T1, taken as the average of three subsequent heart evolutions and measured separately for each lead. Only cases in which ECG waveform without significant artifact or interferences was obtained in at least 8 leads in both T0 and T1 will be analyzed.

From the obtained values, the P wave dispersion will be calculated (as the difference in the length of the P wave in two leads in which the average time of three evolutions was the longest and the shortest) and the PQ dispersion (as the difference in the length of the PQ interval in two leads in which the average time of three evolutions was the longest and the shortest). The obtained data will be subjected to statistical analysis taking into account the side of the body on which the intervention was performed.

ELIGIBILITY:
Inclusion Criteria:

* woman above 18 years of age, legally able of giving informed consent
* participants previously qualified for elective breast surgery due to neoplasm, with or without axillary node dissection
* physical status corresponding to class I or II in American Society of Anaesthesiologist classification

Exclusion Criteria:

* lack of consent to participation or to regional anaesthesia for planned surgery
* bilateral operation planned
* symptomatic circulatory disease at the time of qualification, artificial heart pacemaker presence, positive history of arrythmia
* allergy to amide local anaesthetics
* severe deformation of thoracic spine
* use of medications with "known" or "possible" potential of QT prolongation, according to Arizona Center for Education and Research on Therapeutics [AZCERT] Inc. list, in 5 days preceding the intervention
* use of beta-adrenolytic medications in 5 days preceding the intervention All exclusion criteria except the last one are based on the original study protocol (NCT05822076).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women above 18 years of age, without severe systemic comorbidities, patients of University Clinical Centre of Medical University of Gdańsk qualified for elective breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
P wave time | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of P wave time (as a mean from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
P wave minimal time | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of shortest P wave time (from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
P wave maximal time | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of longest P wave time (from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
PR interval | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of PR interval (as a mean from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
PR minimal interval | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of PR minimal interval (from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
PR maximal interval | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of PR maximal interval (from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]

SECONDARY OUTCOMES:
P wave dispersion | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of P wave dispersion (calculated as a difference between the longest and shortest P wave time from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
P wave index | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference of standard deviations from P wave durations (from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]
PR interval dispersion | from 6 up to 15 minutes (according to time of developement of sufficient block distribution)
  difference in milliseconds of PR interval dispersion (calculated as a difference between the longest and shortest PR interval from all measured leads) between baseline ECG [T0] and ECG after confirmation of sufficient area of sensory block [T1]

CONTACTS AND LOCATIONS:
Locations (1):
- Gdański Uniwersytet Medyczny, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided